CLINICAL TRIAL: NCT04493944
Title: Edible Seaweeds and Health: Quality Biomarkers to Support Consumer Acceptance
Acronym: (CuisiAlg)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Laval University (Other)
Collaborators: Quebec Maritime Network (Odyssee Saint-Laurent) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2020-016/11-02-2020
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Food Habits; Self Efficacy
Keywords: Seaweeds, Food skills, Self Efficacy
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (with culinary workshop) (Experimental): This group will be composed of participants that will answer online questionnaires before and after the study, and will participate in a culinary workshop with a chef (3 hours).
  Interventions: Behavioral: Culinary workshop
- Control group (without culinary workshop) (No Intervention): This group will be composed of participants that will answer online questionnaires before and after the study.

INTERVENTIONS:
Behavioral: Culinary workshop — A 3-hour culinary workshop will be led by a chef. The aim of this workshop will be to develop participants' culinary skills related to the preparation and consumption of recipes based on seaweeds, through various practical activities in the kitchen (starter, main course, dessert). An evaluation questionnaire will be completed at the end of the workshop.
  Arms: Intervention group (with culinary workshop)

SUMMARY:
Seaweeds have been part of the diet of Asian countries for thousands of years, but consumption by Quebecers remains unfamiliar. Because of their rich nutrients content and unique bioactive compounds, seaweeds have a great dietary potential. The overall objective of the project is to determine the potential for sustainable local exploitation of St. Lawrence seaweeds by assessing their quality under growing conditions and following processing, and to use them as a basis for culinary innovations for both industry and consumers. Our specific objectives are as follows:

1. To assess the impact of environmental factors on the specific profile of biomarkers of nutritional quality and health potential of harvested or cultivated seaweed;
2. To determine the impact of processing on the profile of biomarkers of nutritional quality and health potential of harvested and cultivated seaweed;
3. To study changes in dietary attitudes and behaviours through a culinary workshop promoting the acceptance of seaweeds and their appropriation as an ingredient by consumers.

The application for ethical approval and this trial registration applies only to Specific Objective 3.

DETAILED DESCRIPTION:
For recruitment purposes, adults interested in cooking and consuming Quebec seaweeds will be randomly assigned to an experimental group (n=16 x 3 groups, ingredients, recipes and a culinary workshop) or a control group (n=16 x 3 groups, ingredients and recipes). Online questionnaires will be administered via the secure platform of INAF (FANI) at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* be interested in cooking and consuming Quebec seaweeds in various forms
* be available to fill out online questionnaires and perhaps participate in a culinary workshop in Quebec City

Exclusion Criteria:

* have allergies and dietary restrictions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Cooking and food-preparation practices with seaweeds | 2 months
  To evaluate the impact of the culinary workshop on cooking practices of participants (self-efficacy, food attitude, food structure). Will be conducted at baseline and at the end of the study.
Consumption of seaweeds | 2 months
  To evaluate the impact of the culinary workshop on consumption of seaweeds by participants. Will be conducted at baseline and at the end of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Provencher, PhD, Principal Investigator — co-investigator, responsible for Specific Objective 3
Locations (1):
- Institue of Nutrition and Functional Foods (INAF), Québec, Quebec, Canada